CLINICAL TRIAL: NCT04066283
Title: Novel Evaluations of Aging and Gender-Affirming Hormone Therapy on Vascular Endothelial Function and Metabolic Profiles in Transgender Women Compared to Age Group-Matched Cisgender Adults
Brief Title: Effects of Aging and Gender-Affirming Hormone Therapy on Vascular Endothelial Function and Metabolic Profiles in Transgender Women
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 18-2258
Record Dates: First submitted 2019-06-17; First posted 2019-08-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Transgender; Gender Identity; Vascular Stiffness; Vascular Inflammation; Insulin Sensitivity; Blood Pressure; Lipid Disorder; Appetitive Behavior
MeSH Terms: conditions — Insulin Resistance; Lipid Metabolism Disorders; Appetitive Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Endothelial cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older transgender women: This cohort will consist of transgender women aged 50-75 years old who have taken estradiol and spironolactone for at least one year.
  Interventions: Other: No intervention
- Younger transgender women: This cohort will consist of transgender women aged 18-40 years old who have taken estradiol and spironolactone for at least one year.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There was no intervention in this study

SUMMARY:
This study will examine markers of vascular endothelial function (vascular health) and metabolic profiles in younger versus older transgender women (people who were assigned male at birth but whose gender identity is female). Data will also be compared to those from cisgender women and men.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years old or 50-75 years old
* Identify as a transgender woman
* Have taken estradiol and spironolactone for at least one year
* Currently taking oral or transdermal estradiol

Exclusion Criteria:

* Don't identify as a transgender woman
* Not currently taking estradiol or spironolactone
* Have been on estradiol and spironolactone for less than one year
* History of orchiectomy
* Current tobacco smoker
* Current illicit drug use
* History of prior or active estrogen-dependent neoplasms
* Acute liver or gallbladder disease
* Venous thromboembolism
* Hypertriglyceridemia >500 mg/dL
* Fasted plasma glucose >7.0 mmol/L or previously treated diabetes
* Resting blood pressure >140/90 mmHg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women (people who were assigned male at birth but whose gender identity is female). They may or may not have legally changed their gender marker.
Study Population: Transgender women from the Denver metropolitan area and/or who utilize health care at University of Colorado Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of endothelial function (flow-mediated dilation (FMD) | Baseline
  Brachial artery flow-mediated dilation (FMD), as measured by ultrasound.

SECONDARY OUTCOMES:
Evaluation of carotid artery compliance | Baseline
  The carotid artery compliance index indicates how elastic the artery is. The index describes the change in arterial blood volume in response to a change in arterial blood pressure. Lower numbers are associated with worse outcomes (less elastic arteries).
Evaluation of carotid artery beta stiffness index | Baseline
  The carotid artery beta stiffness index indicates how stiff the artery is. Higher numbers are associated with worse outcomes (stiffer artery).
Carotid artery intimal-medial thickness | Baseline
Evaluation of oxidant burden: oxidized LDL | Baseline
  Oxidized low-density lipoprotein (LDL) measured in the blood and endothelial cells.
Evaluation of oxidant burden: nitrotyrosine | Baseline
  Nitrotyrosine measured in the blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: NFkB | Baseline
  Protein NFkB (nuclear factor kappa-light-chain-enhancer of activated B cells) measured in blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: MCP-1 | Baseline
  Monocyte Chemoattractant Protein-1 (MCP-1) measured in blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: IL-6 | Baseline
  Interleukin 6 (IL-6) measured in blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: CRP | Baseline
  C-reactive protein (CRP) measured in blood and endothelial cells.
Blood pressure | Baseline
Plasma lipid concentrations: total cholesterol | Baseline
  Total cholesterol will be determined at baseline.
Plasma lipid concentrations: triglycerides | Baseline
  Triglycerides will be determined at baseline.
Insulin sensitivity | Baseline
Whole body composition: Percent Lean Mass | Baseline
  Percent lean mass will be determined using dual energy x-ray absorptiometry.
Whole body composition: Percent Fat Mass | Baseline
  Percent fat mass will be determined using dual energy x-ray absorptiometry.
Regional body composition: Percent Lean Mass | Baseline
  Regional percent lean mass will be determined using dual energy x-ray absorptiometry.
Regional body composition: Percent Fat Mass | Baseline
  Regional percent fat mass will be determined using dual energy x-ray absorptiometry.
Weight changes | Baseline
Appetite ratings | Baseline
Appetite-related peptides | Baseline
D-Dimer | Baseline
Alcohol use | Baseline
Depression symptoms | Baseline
Physical activity monitoring | 7 days
  Physical activity will me monitored for 7 days with an ActivPALmonitor
Energy intake | 3 days
  Energy intake will be estimated with a 3-day food diary

CONTACTS AND LOCATIONS:
Overall Officials: Sean Iwamoto, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No